CLINICAL TRIAL: NCT03653325
Title: Can Non-invasive Multi-wavelength Monitoring of Out of Hospital Cardiac Arrest Having a Sustained ROSC Reduce Hyperoxia and Hypoxia During Hospital Transfer
Brief Title: ORI to Reduce Hyperoxia After Out Hospital Cardiac Arrest
Acronym: ORI-ONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Collaborators: Centre Hospitalier Universitaire Brugmann (Other); Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORI one
Record Dates: First submitted 2018-07-17; First posted 2018-08-31 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Oxygen Toxicity
Keywords: hyperoxia; post rosc; oxygen reserve index; Fi02 titration; post cardiac arrest care; oxygen
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Hyperoxia | interventions — Oximetry

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- interventional arm (Experimental): In the interventional arm of the study clinicians will be encouraged to titrate oxygen FiO2 according to the following table:
  Interventional arm (FiO2 adaptation every 2-3 min) :
  ORI >0.5 and SatO2>98% and FiO2>0.5 FiO2 reduction of 0.2 ORI>0.01 and ORI<0.5 and SatO2>98% and FiO2>0.5 FiO2 reduction of 0.1 ORI >0.5 and SatO2>98% and FiO2≤0.5 FiO2 reduction of 0.1 ORI>0.01 and ORI<0.5 and SatO2>98% and FiO2≤0.5 FiO2 reduction of 0.05 ORI=0 et SatO2 94 - 98% no modification of FiO2 SatO2<94% + SatO2> 90% increase FiO2 by 0.05 SatO2<90% and SatO2>86 increase FiO2 by 0.1 SatO2<86% and SatO2> 80% increase FiO2 by 0.2 SatO2<80% FiO2 at 1
  In the absence of a ORI measurement reading FiO2 will be adapted as in the observational arm according to SatO2 only.
  Interventions: Device: ORI measurement; Device: oxygen saturation measurement
- Observational arm (Active Comparator): Observational arm (adaptation every 2-3 min):
  oxygen saturation measurement SatO2>98% and FiO2>0.5 reduction of FiO2 by 0.1 SatO2>98% and FiO2≤0.5 reduction of FiO2 by 0.05 SatO2 94 - 98% no modification of FiO2 SatO2<94% + SatO2> 90% increase FiO2 by 0.05 SatO2<90% and SatO2>86 increase FiO2 by 0.1 SatO2<86% and SatO2> 80% increase FiO2 by 0.2 SatO2<80% FiO2 at 1
  Interventions: Device: oxygen saturation measurement

INTERVENTIONS:
Device: ORI measurement — Oxygen (FiO2) will be titrated according to ORI index and Oxygen saturation.
  Arms: interventional arm
Device: oxygen saturation measurement — Oxygen (FiO2) will be titrated according to oxygen saturation

SUMMARY:
The investigator's research proposal is a randomized controlled study evaluating two different monitoring strategies to titrate FiO2 in order to rapidly and safely achieve optimal SatO2 targets during early ROSC of non-traumatic OHCA in adults.

Primary hypothesis:

Monitoring transport to hospital of sustained ROSC of OHCA patients using multiple wavelength detectors that allow ORI continuous measurement will reduce hyperoxia and hypoxia burden associated with transport.

Secondary hypothesis:

Multiple wavelength detectors allowing ORI continuous measurement will reduce hyperoxia at ER admission as measured via blood gas analysis.

Tertiary study hypothesis:

Multiple wavelength detectors allowing ORI continuous measurement will reduce reperfusion neuronal injury measured through NSE levels at 48h post ROSC

DETAILED DESCRIPTION:
Oxygen has a pivotal role in emergency medicine as a lifesaving therapy in numerous situations. In order to avoid hypoxia-related morbidity and mortality, oxygen is delivered in emergencies in a liberal way, even when hypoxia is not confirmed. Nevertheless, as every medication, experimental and clinical studies have highlighted potential side effects of high oxygen tension that could worsen outcome. Cardiac arrest is the archetypal situation given the urgent need of rapid oxygen delivery to organs. However, this global ischemia-reperfusion syndrome produces high amounts ROS that could magnify the damages of the ischemic period and might be significantly increased by high oxygen tension. Thus, hyperoxia in the post-resuscitation context of cardiac arrest is an important topic. Advances in noninvasive oxygen monitoring can now allow for non-invasive monitoring of hyperoxia in pre-hospital settings. So far, despite the recognized urgent need for advancements in the management of oxygen delivery during early ROSC, studies have been exclusively retrospective and interventional studies failed to safely titrate oxygen in the prehospital context possibly due to lack of technological support7. The aim of investigator's is therefore to determine whether technological advances can allow for a safer and more accurate delivery of oxygen in the early ROSC of OHCA, reducing ROS damage. Further research should then, if our hypothesis would be confirmed, reproduce the data in different settings and further investigate whether better oxygen administration during early ROSC improves patients' outcome.

Patient showing a sustained ROSC after an OHCA will be monitored according to current hospital protocols during pre-hospital transport. In addition to traditional monitoring patients will all be monitored with a Masimo device allowing continuous non-invasive measurement of ORI. Patients will be randomly assigned to blinded measurement of ORI (not allowing the clinician to visualize collected information through additional monitoring) or bi-modal monitoring (allowing the clinician to gather information both form traditional monitoring and from additional monitoring showing ORI values). In the latter case clinicians participant will be encouraged to target an ORI lower than 0.5 together with a SatO2>91%. In case of blinded measurement of ORI clinicians will manage ventilation according to standard SatO2 targets (94-98%). Ventilator settings in both groups will be managed in order to target an end-tidal CO2 (ETCO2) between 35 and 45mmHg.

An arterial blood sample and a central body temperature will be taken at hospital admission.

The arterial blood sample will be analysed for glucose, pH, PaCO2 and PaO2 and corrected for temperature in order to calculate dissolved oxygen.

A second blood sample will be done at 48h to measure NSE. A standardised form will be filled by the pre-hospital physician participant gathering information about no flow time, low flow time, first assessed rhythm, BMI, smoking habit and patient demographics.

ELIGIBILITY:
Inclusion Criteria:

* out hospital cardiac arrest
* non traumatic etiology
* ROSC achieved

Exclusion Criteria:

* less 18 year
* traumatic etiology
* prisonnier
* pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
normoxia index | at date of randomisation, from Time of randomisation at ROSC up to time of hospital admission.
  Normoxia index = 1- ( Hypoxia index + Hyperoxia index). Varies from 0 to 1. 1 being a patient without hyper or hypoxia at any moment.
  Hypoxia index=the area above the curve of SatO2 normalized on time. Varies from 0 to 1. 1 being a patient hypoxic during all experiment.
  Hyperoxia index=the area below the curve of ORI measurements and the arbitrary lower limit of an ORI index of 0 representing a PaO2 of approximatively 80mmHg. Varies from 0 to 1. 1 being a patient hyperoxic during all experiment.

SECONDARY OUTCOMES:
Dissolved Oxygen in admission Blood gas sample (DO) | at date of randomisation from time of hospital admission up to 30 minutes after time of hospital admission
  DO=Kh x PaO2. Range are expected to be from 0 to 6. 6 is associating with a higher hyperoxia.
PaO2 in admission blood gas sample | at date of randomisation from time of hospital admission up to 30 minutes after time of hospital admission
  PaO2 as from arterial blood sample. Range expected to be from 20mmHg to 600mmHg. Values between 60mmHg to 150mmHg being associated with the best prognosis

OTHER OUTCOMES:
NSE concentrations | 48 hours after ROSC
  NSE concentrations as from laboratory measurements, biomarker of neuronal damage. Range are expected from 0,15µg/L up to 350 µg/L/ The highest is the result, the worst is the prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: stefano Malinverni, Principal Investigator — Centre Hospitalier Universitaire Saint Pierre
Locations (2):
- Belgium (2):
  - CHU Saint Pierre, Brussels
  - Centre Hospitalier Universitaire Brugmann, Brussels

IPD SHARING:
Plan to Share IPD: Yes
After publication all IPD inherent with the publication will be made available through the researchgate.com profile of the principal investigator
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After publication
Access Criteria: Access will be granted to any researcher requesting access through Researchgate.com

REFERENCES:
- [Derived] Malinverni S, Wilmin S, Stoll T, de Longueville D, Preseau T, Mohler A, Bouazza FZ, Annoni F, Gerard L, Denoel P, Boutrika I. Postresuscitation oxygen reserve index-guided oxygen titration in out-of-hospital cardiac arrest survivors: A randomised controlled trial. Resuscitation. 2024 Jan;194:110005. doi: 10.1016/j.resuscitation.2023.110005. Epub 2023 Oct 18. PMID 37863418